CLINICAL TRIAL: NCT04462445
Title: Prospective Translational Study Investigating Possible Molecular prEdictors of Resistance to First-Line pazopanIb in Metastatic reNal Cell Carcinoma
Brief Title: Prospective Translational Study Investigating Possible Molecular prEdictors of Resistance to First-Line pazopanIb
Acronym: PIPELINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 146-14
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-06

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pazopanib (Experimental): Pazopanib 800 mg (2x400mg ) taken orally daily as per clinical practice
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib

SUMMARY:
This is a prospective, single-arm, monocentric translational study designed to evaluate possible biomarkers of resistance to the first line of therapy with pazopanib in patients with metastatic renal cell carcinoma (mRCC) who have not received systemic therapy in both the adjuvant and metastatic phases.

DETAILED DESCRIPTION:
a prospective, single-arm, monocentric translational study

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Unresectable advanced or metastatic renal cell carcinoma (RCC) with component of clear cell histology and/or component of sarcomatoid histology that has not been previously treated with any systemic agent, including treatment in the adjuvant setting
* Availability of a representative formalin-fixed paraffin-embedded fractional Fokker-Planck equation (FFPE) tumor specimen collected within 24 months of starting first-line pazopanib that enables the definitive diagnosis of renal cell carcinoma (RCC) (the archival specimen must contain adequate viable tumor tissue to enable candidate biomarkers status; the specimen may consist of a tissue block or at least 15 unstained serial sections; for core needle biopsy specimens at least two cores should be available for evaluation)
* Measurable disease as defined by RECIST v1.1
* Age ≥18 years

Hematology Absolute neutrophil count (ANC)≥1.5 X 109/L Hemoglobin ≥9 g/dL (5.6 mmol/L) Platelets ≥100 X 109/L Prothrombin time (PT) or international normalized ratio (INR)b ≤1.5 X upper limit of normal (ULN) Activated partial thromboplastin time (aPTT) ≤1.5 X upper limit of normal (ULN) Hepatic Total bilirubin ≤1.5 X upper limit of normal (ULN) Alanine amino transferase (ALT) and Aspartate aminotransferase (AST)c 2.5 X upper limit of normal (ULN) Patients with documented liver metastases <5 X upper limit of normal (ULN) Renal Serum creatinine 1.5 mg/dL (133 µmol/L) Or, if >1.5 mg/dL: Calculated creatinine clearance (ClCR) (reference appropriate appendix) ≥30 mL/min to ≥ 50 mL/min Urine Protein to Creatinine Ratio (UPC; appropriate appendix)<1 Or, 24-hour urine protein <1g

- Eastern Cooperative Oncology Group (ECOG) performance Status 0-1

Exclusion Criteria:

* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to: active peptic ulcer disease, known intraluminal metastatic lesion/s with risk of bleeding, inflammatory bowel disease (e.g. ulcerative colitis, Chrohn's disease), or other gastrointestinal conditions with increased risk of perforation, history of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
* History of any one or more of the following cardiovascular conditions within the past 6 months:

cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA) - Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 millimetre (s) of mercury (mmHg) or diastolic blood pressure (DBP) of ≥ 90 millimetre (s) of mercury (mmHg)].

Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals. At least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and BP measurement. These three values should be averaged to obtain the mean diastolic blood pressure and the mean systolic blood pressure. The mean SBP / DBP ratio must be <140/90 millimetre (s) of mercury (mmHg) (OR 150/90 millimetre (s) of mercury (mm Hg), if this criterion is approved by Safety Review Team) in order for a subject to be eligible for the study

- History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible

* Major surgery or trauma within 28 days prior to first dose of pazopanib and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage Note: Lesions infiltrating major pulmonary vessels (contiguous tumour and vessels) are excluded; however, the presence of a tumor that is touching, but not infiltrating (abutting) the vessels is acceptable (CT with contrast is strongly recommended to evaluate such lesions).
* Large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed.
* Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of the bronchi are allowed.
* Recent hemoptysis (½ teaspoon of red blood within 8 weeks before first dose of study drug).
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Treatment with any of the following anti-cancer therapies:
* chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of Pazopanib

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
A panel of possible predictive candidate biomarkers of resistance to anti-angiogenic targeted tyrosine kinase inhibitor (TKI) | 18 months
  using next-generation sequencing (NGS) methods for future research. This will be done by within-patient comparison of metastatic tissue samples taken on commencement of first-line pazopanib, and secondly on development of TKI resistance
The Overall Response Rate (ORR) | 18 months
  evaluate per RECIST v.1.1 criteria in mRCC patients treated with first-line pazopanib in order to either correlate circulating angiogenic factors (CAFs) levels and gene candidate biomarkers status to clinical outcome when resistance develops

SECONDARY OUTCOMES:
Identification of other protein markers circulating in blood, | 18 months
  To obtain serial blood samples from patients whilst they are being treated with pazopanib
compare the frequency of previously defined promising circulating predictive biomarkers for pazopanib treatment | 18 months
  between blood samples taken at commencement of therapy (baseline) and at the time of progressive disease (PD) as per RECIST 1.1 criteria as well as changes of interleukin 8 (IL-8), c-Met and hematopoietic growth factor (HGF) expression between metastatic tumour tissue samples in order to better understand changes in the tumor and in the levels of circulating angiogenic factors as resistance develops.
Collect Data | 18 months
  prospective and retrospective demographic, clinical and pathological data on patients who enter the study, enabling current and future correlation of biomarkers to clinical outcomes
Perform subgroup analyses | 18 months
  comparing the tissue and blood biomarkers identified in patients who developed secondary resistance with those biomarkers identified in patients who have primary resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI

REFERENCES:
- [Result] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Result] Motzer RJ, Bander NH, Nanus DM. Renal-cell carcinoma. N Engl J Med. 1996 Sep 19;335(12):865-75. doi: 10.1056/NEJM199609193351207. No abstract available. PMID 8778606
- [Result] Latif F, Tory K, Gnarra J, Yao M, Duh FM, Orcutt ML, Stackhouse T, Kuzmin I, Modi W, Geil L, et al. Identification of the von Hippel-Lindau disease tumor suppressor gene. Science. 1993 May 28;260(5112):1317-20. doi: 10.1126/science.8493574.
- [Result] George DJ, Kaelin WG Jr. The von Hippel-Lindau protein, vascular endothelial growth factor, and kidney cancer. N Engl J Med. 2003 Jul 31;349(5):419-21. doi: 10.1056/NEJMp030061. No abstract available. PMID 12890838
- [Result] Schwandt A, Wood LS, Rini B, Dreicer R. Management of side effects associated with sunitinib therapy for patients with renal cell carcinoma. Onco Targets Ther. 2009 Feb 18;2:51-61. doi: 10.2147/ott.s4052. PMID 20616894
- [Result] Sonpavde G, Hutson TE, Sternberg CN. Pazopanib, a potent orally administered small-molecule multitargeted tyrosine kinase inhibitor for renal cell carcinoma. Expert Opin Investig Drugs. 2008 Feb;17(2):253-61. doi: 10.1517/13543784.17.2.253. PMID 18230058
- [Result] Kumar R, Crouthamel MC, Rominger DH, Gontarek RR, Tummino PJ, Levin RA, King AG. Myelosuppression and kinase selectivity of multikinase angiogenesis inhibitors. Br J Cancer. 2009 Nov 17;101(10):1717-23. doi: 10.1038/sj.bjc.6605366. Epub 2009 Oct 20. PMID 19844230
- [Result] Sternberg CN, Davis ID, Mardiak J, Szczylik C, Lee E, Wagstaff J, Barrios CH, Salman P, Gladkov OA, Kavina A, Zarba JJ, Chen M, McCann L, Pandite L, Roychowdhury DF, Hawkins RE. Pazopanib in locally advanced or metastatic renal cell carcinoma: results of a randomized phase III trial. J Clin Oncol. 2010 Feb 20;28(6):1061-8. doi: 10.1200/JCO.2009.23.9764. Epub 2010 Jan 25. PMID 20100962
- [Result] Motzer RJ, Hutson TE, Cella D, Reeves J, Hawkins R, Guo J, Nathan P, Staehler M, de Souza P, Merchan JR, Boleti E, Fife K, Jin J, Jones R, Uemura H, De Giorgi U, Harmenberg U, Wang J, Sternberg CN, Deen K, McCann L, Hackshaw MD, Crescenzo R, Pandite LN, Choueiri TK. Pazopanib versus sunitinib in metastatic renal-cell carcinoma. N Engl J Med. 2013 Aug 22;369(8):722-31. doi: 10.1056/NEJMoa1303989. PMID 23964934
- [Result] Escudier B, Porta C, Bono P, Powles T, Eisen T, Sternberg CN, Gschwend JE, De Giorgi U, Parikh O, Hawkins R, Sevin E, Negrier S, Khan S, Diaz J, Redhu S, Mehmud F, Cella D. Randomized, controlled, double-blind, cross-over trial assessing treatment preference for pazopanib versus sunitinib in patients with metastatic renal cell carcinoma: PISCES Study. J Clin Oncol. 2014 May 10;32(14):1412-8. doi: 10.1200/JCO.2013.50.8267. Epub 2014 Mar 31. PMID 24687826
- [Result] Ravaud A, Gross-Goupil M. Overcoming resistance to tyrosine kinase inhibitors in renal cell carcinoma. Cancer Treat Rev. 2012 Dec;38(8):996-1003. doi: 10.1016/j.ctrv.2012.01.003. Epub 2012 Feb 12. PMID 22330762
- [Result] Hutson TE. Targeted therapies for the treatment of metastatic renal cell carcinoma: clinical evidence. Oncologist. 2011;16 Suppl 2(Suppl 2):14-22. doi: 10.1634/theoncologist.2011-S2-14. PMID 21346036
- [Result] Hernandez-Yanez M, Heymach JV, Zurita AJ. Circulating biomarkers in advanced renal cell carcinoma: clinical applications. Curr Oncol Rep. 2012 Jun;14(3):221-9. doi: 10.1007/s11912-012-0231-2. PMID 22434312
- [Result] Bergers G, Hanahan D. Modes of resistance to anti-angiogenic therapy. Nat Rev Cancer. 2008 Aug;8(8):592-603. doi: 10.1038/nrc2442. PMID 18650835
- [Result] Shojaei F, Lee JH, Simmons BH, Wong A, Esparza CO, Plumlee PA, Feng J, Stewart AE, Hu-Lowe DD, Christensen JG. HGF/c-Met acts as an alternative angiogenic pathway in sunitinib-resistant tumors. Cancer Res. 2010 Dec 15;70(24):10090-100. doi: 10.1158/0008-5472.CAN-10-0489. Epub 2010 Oct 15. PMID 20952508
- [Result] Birchmeier C, Birchmeier W, Gherardi E, Vande Woude GF. Met, metastasis, motility and more. Nat Rev Mol Cell Biol. 2003 Dec;4(12):915-25. doi: 10.1038/nrm1261. No abstract available. PMID 14685170
- [Result] Zhang YW, Su Y, Volpert OV, Vande Woude GF. Hepatocyte growth factor/scatter factor mediates angiogenesis through positive VEGF and negative thrombospondin 1 regulation. Proc Natl Acad Sci U S A. 2003 Oct 28;100(22):12718-23. doi: 10.1073/pnas.2135113100. Epub 2003 Oct 10. PMID 14555767
- [Result] Waugh DJ, Wilson C. The interleukin-8 pathway in cancer. Clin Cancer Res. 2008 Nov 1;14(21):6735-41. doi: 10.1158/1078-0432.CCR-07-4843. PMID 18980965
- [Result] Mizukami Y, Jo WS, Duerr EM, Gala M, Li J, Zhang X, Zimmer MA, Iliopoulos O, Zukerberg LR, Kohgo Y, Lynch MP, Rueda BR, Chung DC. Induction of interleukin-8 preserves the angiogenic response in HIF-1alpha-deficient colon cancer cells. Nat Med. 2005 Sep;11(9):992-7. doi: 10.1038/nm1294. Epub 2005 Aug 28. PMID 16127434
- [Result] Huang D, Ding Y, Zhou M, Rini BI, Petillo D, Qian CN, Kahnoski R, Futreal PA, Furge KA, Teh BT. Interleukin-8 mediates resistance to antiangiogenic agent sunitinib in renal cell carcinoma. Cancer Res. 2010 Feb 1;70(3):1063-71. doi: 10.1158/0008-5472.CAN-09-3965. Epub 2010 Jan 26. PMID 20103651
- [Result] Kapur P, Pena-Llopis S, Christie A, Zhrebker L, Pavia-Jimenez A, Rathmell WK, Xie XJ, Brugarolas J. Effects on survival of BAP1 and PBRM1 mutations in sporadic clear-cell renal-cell carcinoma: a retrospective analysis with independent validation. Lancet Oncol. 2013 Feb;14(2):159-167. doi: 10.1016/S1470-2045(12)70584-3. Epub 2013 Jan 16. PMID 23333114
- [Result] Jorgensen TJ, Ruczinski I, Kessing B, Smith MW, Shugart YY, Alberg AJ. Hypothesis-driven candidate gene association studies: practical design and analytical considerations. Am J Epidemiol. 2009 Oct 15;170(8):986-93. doi: 10.1093/aje/kwp242. Epub 2009 Sep 17. PMID 19762372
- [Result] Tran HT, Liu Y, Zurita AJ, Lin Y, Baker-Neblett KL, Martin AM, Figlin RA, Hutson TE, Sternberg CN, Amado RG, Pandite LN, Heymach JV. Prognostic or predictive plasma cytokines and angiogenic factors for patients treated with pazopanib for metastatic renal-cell cancer: a retrospective analysis of phase 2 and phase 3 trials. Lancet Oncol. 2012 Aug;13(8):827-37. doi: 10.1016/S1470-2045(12)70241-3. Epub 2012 Jul 2. PMID 22759480
- [Result] Galluzzi L, Buque A, Kepp O, Zitvogel L, Kroemer G. Immunological Effects of Conventional Chemotherapy and Targeted Anticancer Agents. Cancer Cell. 2015 Dec 14;28(6):690-714. doi: 10.1016/j.ccell.2015.10.012. PMID 26678337
- [Result] Donini M, Buti S, Lazzarelli S, Bozzetti R, Rivoltini L, Camisaschi C, Castelli C, Bearz A, Simonelli C, Lo Re G, Mattioli R, Caminiti C, Passalacqua R; GOIRC (Italian Oncology Group for Clinical Research). Dose-finding/phase II trial: bevacizumab, immunotherapy, and chemotherapy (BIC) in metastatic renal cell cancer (mRCC). Antitumor effects and variations of circulating T regulatory cells (Treg). Target Oncol. 2015 Jun;10(2):277-86. doi: 10.1007/s11523-014-0337-6. Epub 2014 Sep 19. PMID 25230695
- [Result] Castelli C, Rivoltini L, Rodolfo M, Tazzari M, Belgiovine C, Allavena P. Modulation of the myeloid compartment of the immune system by angiogenic- and kinase inhibitor-targeted anti-cancer therapies. Cancer Immunol Immunother. 2015 Jan;64(1):83-9. doi: 10.1007/s00262-014-1576-1. Epub 2014 Jul 4. PMID 24993564